CLINICAL TRIAL: NCT04550949
Title: A Multi-center, Randomized, Double-blind, Comparative Study to Evaluate the Clinical Efficacy and Safety of QL1206 and Xgeva® in Patients With Bone Metastases From Solid Tumors
Brief Title: To Evaluate the Efficacy and Safety of QL1206 and Xgeva in Patients With Bone Metastases From Solid Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1206-003
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Bone Metastases
MeSH Terms: interventions — QL1206; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1206 (Experimental): QL1206 injection(120mg)was administered subcutaneously once every 4 weeks for a maximum of 13 consecutive doses throughout the trial, according to the investigator's assessment.
  Interventions: Drug: QL1206
- Xgeva® (Active Comparator): Xgeva® injection(120mg) was administered subcutaneously every 4 weeks for a maximum of 13 cumulative doses throughout the trial,according to the investigator's assessment.
  Interventions: Drug: Xgeva

INTERVENTIONS:
Drug: QL1206 — The active ingredient of QL1206 is a recombinant human anti-RANKL monoclonal antibody ,subcutaneous injection of 120 mg (1.7ml)every 4 weeks for a maximum of 13 consecutive doses throughout the trial.
  Other Names: recombinant human anti-RANKL monoclonal antibody injection
  Arms: QL1206
Drug: Xgeva — The active ingredient of Xgeva® is denosumab,subcutaneous injection of 120 mg (1.7ml)every 4 weeks for a maximum of 13 consecutive doses throughout the trial.
  Other Names: Denosumab Injection
  Arms: Xgeva®

SUMMARY:
A multi-center, randomized, double-blind, comparative study to evaluate the clinical efficacy and safety of QL1206 and Xgeva® in patients with bone metastases from solid tumors.

DETAILED DESCRIPTION:
This is A multi-center, randomized, double-blind, comparative clinical trial.

The primary objective is to evaluate whether the clinical efficacy of QL1206 and Xgeva® are similar in patients with bone metastases from solid tumors.

The secondary objective are to evaluate whether the clinical safety and immunogenicity of QL1206 and Xgeva® are similar in patients with bone metastases from solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Through the explanation of the researcher or the researcher's authorized representative, the subject has understood the nature and purpose of the study, as well as the research procedure, and the subject has signed the written informed consent;
2. Radiologic evidence (i.e. X-ray examination, computed tomography CT, magnetic resonance imaging MRI, positron emission computed tomography PET-CT) in grade III grade A hospitals has been documented (within 3 months prior to study administration) that there is at least one bone metastasis;
3. The ECOG score was 0-2.
4. Chinese adults with solid tumor confirmed by histological or cytological examination (age ≥18 years, ≤80 years).

Exclusion Criteria:

1. Patients who had received any kind of intravenous or oral bisphosphonates before administration of the first study drug (those who had previously used an intravenous or oral bisphosphonates but had a continuous use time of less than 3 months and more than 5 years before the administration of this study could be included in the study).
2. Previous treatment with denosumab.
3. Previous or ongoing osteomyelitis or osteonecrosis of the jaw ONJ , active dental disease or jaw bone disease requiring oral surgery, the wound of dental operation or oral surgery has not healed well, or invasive dental operation has been planned during the study period.
4. Plan to perform radiotherapy or or bone surgery. Patients who received radiotherapy within one month before the first study drug administration were not allowed to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
uNTx/uCr | from baseline to week 13
  Compare QL1206 and Xgeva® for percentage change in bone conversion index (BTM) - urinary type I collagen cross-linked peptide (uNTx) adjusted for urinary creatinine (uCr) in Chinese subjects with solid tumor bone metastasis (uNTx/uCr from baseline to week 13)

SECONDARY OUTCOMES:
uNTx/uCr | from baseline to weeks 25 and 53
  Compare the percentage change in QL1206 and Xgeva® for bone conversion indicator uNTx/uCr among subjects with solid tumor metastasis (from baseline to weeks 25 and 53).
S-BALP | from baseline to weeks 13, 25, and 53
  Compare the changes of bone specific alkaline phosphatase (S-BALP) from baseline to weeks 13, 25, and 53.
SRE | from baseline to weeks 53
  SRE occurrence

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong

REFERENCES:
- [Derived] Liu Y, Zhang R, Wang X, Di L, Chen Z, Wang J, Sun T, Li Q, Cheng J, Zhang Q, Wang X, Wang J, Gu K, Wei S, Zhang S, Wang X, Sun P, Hao C, Zang A, Li Y, Han C, Kang X, Li Y, Li H. Comparison of efficacy and safety of a proposed biosimilar QL1206 with reference denosumab in patients with bone metastasis from breast cancer: A subgroup analysis of a randomized, double-blinded phase III study. Chin J Cancer Res. 2025 Jun 30;37(3):337-351. doi: 10.21147/j.issn.1000-9604.2025.03.04. PMID 40642487
- [Derived] Li H, Huang Y, Chen Z, Zeng A, Zhang H, Yu Y, Wei S, Li Q, Wang X, Wang X, Wang X, Yang R, Dai X, Bi M, Sun T, Zhang Q, Han C, Li Y, Kang X, Liu Y, Zhang L. Efficacy and Safety of Denosumab Biosimilar QL1206 Versus Denosumab in Patients with Bone Metastases from Solid Tumors: A Randomized Phase III Trial. BioDrugs. 2023 Mar;37(2):259-269. doi: 10.1007/s40259-023-00579-5. Epub 2023 Feb 21. PMID 36802320